CLINICAL TRIAL: NCT06643533
Title: Safety and Efficacy of Fecal Microbiota Transplantation in Reversing Drug Resistance in Patients With Intermediate-advanced Unresectable Hepatocellular Carcinoma Undergoing Transcatheter Arterial Chemoembolization Combined With Lenvatinib Plus Sintilimab.
Brief Title: Fecal Microbiota Transplantation in Reversing Drug Resistance in Unresectable HCC (TALENP004)
Status: Not yet recruiting | Type: Observational
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Mao-Lin Yan, Principal Investigator, Fujian Provincial Hospital
Other Study IDs: TALENP004
Record Dates: First submitted 2024-10-11; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Fecal Microbiota Transplantation; Hepatocellular Carcinoma; TACE; Lenvatinib; PD-1 inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FMT-Resistant HCC Cohort: The triple therapy consists of:
  Transarterial Chemoembolization (TACE): This procedure will be performed every 4-6 weeks based on the presence of significant arterial blood supply to the tumor, with a maximum of 4 TACE treatments allowed.
  Lenvatinib: The generic name of the drug is lenvatinib. It will be administered orally in a dosage of 12mg per day for patients weighing 60kg or more, and 8mg per day for patients weighing less than 60kg. The treatment will be continuous with a fixed daily dosing schedule.
  Sintilimab: It will be given every 3 weeks (Q3W). Fecal Microbiota Transplantation (FMT): The FMT capsules will be prepared by matching the gut microbiome profiles of healthy donors with those of patients who achieved a complete response to the triple therapy. The FMT capsules will be taken orally at a dosage of 30 capsules per day for the first 3 days of each treatment cycle.
  The FMT intervention will be administered in 6 cycles, with each cycle lasting for 21 days (Q3W).
  Interventions: Other: Fecal Microbiota Transplantation

INTERVENTIONS:
Other: Fecal Microbiota Transplantation — The FMT capsules will be prepared by matching the gut microbiome profiles of healthy donors with those of patients who achieved a complete response to the triple therapy. The FMT capsules will be taken orally at a dosage of 30 capsules per day for the first 3 days of each treatment cycle. The FMT intervention will be administered in 6 cycles, with each cycle lasting for 21 days (Q3W). The duration of the treatment will be determined by the response to therapy, with a maximum of 6 cycles or until disease progression, intolerable toxicity, or participant withdrawal of consent. The FMT capsules are intended to modify the gut microbiome to reverse the resistance to the triple therapy and enhance the therapeutic response.

SUMMARY:
This study aims to evaluate the safety and efficacy of fecal microbiota transplantation (FMT) in reversing drug resistance to the triple therapy regimen in patients with unresectable hepatocellular carcinoma (HCC). The triple therapy consists of transarterial chemoembolization (TACE), lenvatinib, and Sintilimab. The study is a prospective, single-arm, multicenter clinical trial involving 15 participants with mid-to-late stage HCC that has progressed despite the triple therapy. FMT capsules will be prepared by matching the gut microbiome profiles of healthy donors to those of patients who achieved complete response (CR) with the triple therapy. The primary endpoints include objective response rate (ORR), treatment-related adverse events (AEs). Secondary endpoints will assess overall survival (OS), progression-free survival (PFS), and disease control rate (DCR), changes in gut microbiome, metabolomics, and immune subsets before and after FMT.

DETAILED DESCRIPTION:
The study is designed to investigate the potential of FMT in overcoming resistance to a combined treatment approach for HCC. The triple therapy under investigation includes TACE, lenvatinib, and a PD-1 inhibitor, which has shown promise in treating HCC but has encountered issues with drug resistance.

This prospective, single-arm, multicenter trial will enroll 15 patients diagnosed with mid-to-late stage HCC that has progressed despite treatment with the triple therapy. The primary objective is to assess the safety and efficacy of FMT in this patient population, with the primary endpoints being ORR, AEs, OS, PFS, and DCR. Secondary endpoints will evaluate the changes in the gut microbiome composition, metabolomic profiles, and immune cell subsets before and after FMT.

Eligible participants must have HCC that has progressed following the triple therapy and meet specific inclusion criteria, including having at least one measurable lesion, an expected survival time greater than three months, and no prior FMT treatment. Exclusion criteria include a history of other malignancies within the past five years, autoimmune diseases, and the use of immunosuppressive agents.

FMT capsules will be made by analyzing the gut microbiome and metabolite profiles of patients who achieved a complete response to the triple therapy, and matching these with healthy donor profiles from a biobank. Patients will receive FMT capsules daily for three days, along with the continuation of the triple therapy. The study will also include procedures for dose adjustments based on adverse events and specific guidelines for managing toxicities related to the study treatments.

The study will conclude with a comprehensive analysis of the primary and secondary endpoints. This trial aims to provide valuable insights into the role of FMT in enhancing the efficacy of cancer treatments and overcoming drug resistance in HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with intermediate to advanced Hepatocellular Carcinoma (HCC) who have experienced disease progression (PD) after treatment with the triple therapy of Transarterial Chemoembolization (TACE), lenvatinib, and sintilimab.
2. Patients must have at least one measurable lesion according to the mRECIST 1.1 criteria (the longest diameter of measurable lesions on CT/MRI scan ≥10mm).
3. Expected survival time greater than 3 months.
4. No prior treatment with Fecal Microbiota Transplantation (FMT).
5. No history of taking probiotics after the diagnosis of HCC.
6. Child-Pugh class A/B.
7. ECOG performance status: ≤1.
8. Age between 18 and 75 years old.
9. No other antitumor treatments except the triple therapy before enrollment.
10. Key organ function indicators meet the following requirements:

    Hematology: Absolute neutrophil count ≥1.5×10^9/L, Hb ≥9.0g/L, Platelets ≥75×10^9/L Liver function: Total bilirubin ≤1.5 times the upper limit of normal (ULN) (≤2.5 times ULN after biliary drainage for obstructive jaundice); Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) ≤5 times ULN, Albumin ≥30g/L Renal function: Serum creatinine ≤1.5mg/dL, Creatinine clearance rate ≥60ml/min Coagulation function: International normalized ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤1.5 times ULN
11. No history of severe arrhythmias, heart failure, severe ventilatory dysfunction, or severe pulmonary infections.
12. Women of childbearing age must agree to use contraceptive measures during the treatment period and for 6 months after the end of treatment, with a negative serum or urine pregnancy test within 7 days before study enrollment, and must not be breastfeeding. Men must agree to use contraceptive measures during the study period and for 6 months after the end of the study.

Exclusion Criteria:

1. Mixed hepatocellular-cholangiocarcinoma.
2. Severe tumor progression (tumor volume occupies two-thirds or more of the liver volume or diffuse intrahepatic lesions).
3. History of allergy to PD-1, lenvatinib, or their components.
4. History of other malignant tumors within the past 5 years, except for cured basal cell carcinoma of the skin, cervical carcinoma in situ, and papillary thyroid cancer.
5. Patients who have undergone organ transplantation or are planning to undergo organ transplantation.
6. Any active autoimmune disease or autoimmune disease with expected recurrence (such as interstitial pneumonia, colitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases and syndromes).
7. History of immunodeficiency; patients who are using immunosuppressants or systemic corticosteroid therapy for immunosuppression and have continued use within 2 weeks before signing the informed consent.
8. Known hereditary or acquired bleeding (such as coagulation disorders) or thrombotic tendencies, such as hemophilia patients; currently using or have recently (within 10 days before the start of the study treatment) used full-dose oral or injectable anticoagulants or thrombolytic drugs for therapeutic purposes (preventive use of low-dose aspirin, low molecular weight heparin is allowed).
9. Serious infections within 4 weeks before enrollment, such as severe pneumonia requiring hospitalization, bacteremia, infectious complications, etc.; baseline chest imaging indicates active pulmonary inflammation, presence of infection symptoms and signs or need for oral or intravenous antibiotic treatment within 2 weeks before the first use of the study drug (excluding the use of antibiotics for prevention).
10. Patients with mental illness; history of abuse of psychotropic drugs, alcoholism, and drug addiction.
11. Chronic intestinal diseases (such as celiac disease, malabsorption, etc.).
12. Pregnant or breastfeeding women.
13. Deemed by the investigator to be unsuitable for participation in this trial for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults aged 18 to 75 with unresectable hepatocellular carcinoma that has progressed after triple therapy, eligible for fecal microbiota transplantation to overcome treatment resistance.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate, ORR | Four weeks after the initiation of medication until the day before surgery
  The Objective response rate (ORR) was defined as the complete response (CR) rate or the partial response (PR) rate according to RECIST1.1.
Adverse events | From the initiation of medication, with recordings made whenever an adverse reaction occurs, assessed up to 12 months
  Grade 1-5 AEs according to NCI-CTCAE V5.0.

SECONDARY OUTCOMES:
Overall survival, OS | From date of enrollment until the date of death from any cause, assessed up to 60 months
  The Overall survival (OS) was defined as the time between receiving treatment and observing death or loss of follow-up for any reason.
Progression free survival, PFS | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  The Progression free survival (PFS) was defined as the time between the start of treatment and the progression of intrahepatic and/or extrahepatic tumors, or the occurrence of death or loss of follow-up for any reason.
Disease control rate, DCR | Four weeks after the initiation of medication until the day before surgery
  The Disease control rate (DCR) was defined as the complete response (CR) rate or the partial response (PR) rate or stable disease (SD) rate according to RECIST1.1.
Gut Microbiome Composition after Fecal Microbiota Transplantation | Baseline and at the end of each treatment cycle (up to 6 cycles)
  The changes in the gut microbiome composition before and after FMT treatment, including diversity and similarity to the donor microbiome.
Gut Microbiome Metabolomic Changes after Fecal Microbiota Transplantation | Baseline and at the end of each treatment cycle (up to 6 cycles)
  The changes in serum and fecal metabolomics before and after FMT.
Gut Microbiome Immune Subset Variations after Fecal Microbiota Transplantation | Baseline and at the end of each treatment cycle (up to 6 cycles)
  The changes in immune cell subsets before and after FMT.

IPD SHARING:
Plan to Share IPD: No